CLINICAL TRIAL: NCT07172841
Title: Randomized Controlled Study on Non-invasive Diagnostics of Shunt Obstruction in Adult Hydrocephalus
Brief Title: Non-invasive Diagnostics of Shunt Obstruction in Adult Hydrocephalus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Department of Neurological Surgery, Sahlgrenska University Hospital (Unknown); Hydrocephalus Research Unit, Sahlgrenska University Hospital (Unknown); Department of Neurological Surgery, Linköping University Hospital (Unknown); Department of Neurology, Linköping University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Dnr 2024-01568-01; Dnr: SU2024-06898 (Other: Biobank Väst)
Record Dates: First submitted 2025-03-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Normal Pressure Hydrocephalus Patients; Normal Pressure Hydrocephalus
Keywords: Volumetry; Shunt obstruction; Shunt patency; NPH; Outcome
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intervention group "Virtual OFF" — Patients randomized to shunt setting "Virtual Off" at the three month follow-up visit. After 5-7 days, the setting will be restored to the previous setting.
Device: Control group (no change in shunt setting) — Patients randomized to continue their shunt setting unchanged

SUMMARY:
The goal of this RCT is to test whether volumetric assessment of magnetic resonance imaging (MRI) could diagnose shunt obstruction in Adult Hydrocephalus patients, and in addition to explore correlations of blood biomarkers surrounding shunt obstruction. Thirdly to investigate correlations with clinical symptom burden before and after surgery.

The main questions it aims to answer are:

Can volumetric assessment of cerebrospinal fluid (CSF) aid in diagnosis of shunt obstruction? Are there dynamical changes in blood biomarker concentrations after shunt obstruction? How are clinical symptom burden and dynamics correlated with blood biomarker changes and volumetric changes in CSF?

After three months of shunt treatment, researchers will compare patients with "Virtual OFF" setting, to explore if simulated shunt obstruction affect measures mentioned above.

Participants randomized to the intervention group will undergo the 'Virtual OFF' setting for a period of 5-7 days, starting 3 months after initiation of shunt treatment. Symptom burden will be assessed preoperatively, at follow-up, and following the week of the shunt setting change. MRI scans will be conducted at these same time points. Participants in the control group will also meet with a nurse, but their shunt settings will remain unchanged. The control group will receive the same symptom assessments and MRI scans as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal pressure hydrocephalus (NPH)
* Treated at either the Hydrocephalus Research Unit in Gothenburg or at the Department of Neurological Surgery at Linköping University Hospital or Sahlgrenska University Hospital

Exclusion Criteria:

* Unable to conform to instructions of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Volumetry of CSF | Preoperatively --> 3 months postop --> 3 months + 5-7 days postop
  Dynamics of volumetric assessment in lateral ventricles and subarachnoid space will be analyzed in groups as a primary outcome measure.

SECONDARY OUTCOMES:
Symptom burden | Preoperatively --> 3 months postop --> 3 months + 5-7 days postop
  Results from 4 clinical tests and 2 self assessment forms will be collected preoperatively, 3 months postop and 3 months + 5-7 days postop. Dynamical changes in symptoms is considered a secondary outcome measure.
  1. Walk-steps: number of steps on a 10 meter walk
  2. Walk-time: number of seconds to walk 10 meters
  3. Color naming test by Stroop
  4. Grooved peg board test
     Self assessment of:
  5. Balance
  6. Urinary continence

OTHER OUTCOMES:
Blood biomarker concentrations | Preoperatively (doctors appointment with diagnostics) --> 1 day preop --> 1 day postop --> 3 months postop --> 3 months + 7 days postop
  Concentrations of biomarkers S100B, GFAP, NFL och Tau will be collected, and their concentration changes could be considered an additional outcome measure.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liden S, Farahmand D, Laurell K. Ventricular volume in relation to lumbar CSF levels of amyloid-beta 1-42, tau and phosphorylated tau in iNPH, is there a dilution effect? Fluids Barriers CNS. 2022 Jul 17;19(1):59. doi: 10.1186/s12987-022-00353-9. PMID 35843939
- [Background] Hallen T, Olsson DS, Hammarstrand C, Farahmand D, Olofsson AC, Jakobsson Ung E, Jakobsson S, Bergquist H, Blennow K, Zetterberg H, Johannsson G, Skoglund T. Circulating brain injury biomarkers increase after endoscopic surgery for pituitary tumors. J Clin Neurosci. 2021 Jul;89:113-121. doi: 10.1016/j.jocn.2021.04.030. Epub 2021 May 12. PMID 34119253
- [Background] Newcombe VFJ, Ashton NJ, Posti JP, Glocker B, Manktelow A, Chatfield DA, Winzeck S, Needham E, Correia MM, Williams GB, Simren J, Takala RSK, Katila AJ, Maanpaa HR, Tallus J, Frantzen J, Blennow K, Tenovuo O, Zetterberg H, Menon DK. Post-acute blood biomarkers and disease progression in traumatic brain injury. Brain. 2022 Jun 30;145(6):2064-2076. doi: 10.1093/brain/awac126. PMID 35377407
- [Background] Saehle T, Farahmand D, Eide PK, Tisell M, Wikkelso C. A randomized controlled dual-center trial on shunt complications in idiopathic normal-pressure hydrocephalus treated with gradually reduced or "fixed" pressure valve settings. J Neurosurg. 2014 Nov;121(5):1257-63. doi: 10.3171/2014.7.JNS14283. Epub 2014 Sep 5. PMID 25192478
- [Background] Farahmand D, Saehle T, Eide PK, Tisell M, Hellstrom P, Wikkelso C. A double-blind randomized trial on the clinical effect of different shunt valve settings in idiopathic normal pressure hydrocephalus. J Neurosurg. 2016 Feb;124(2):359-67. doi: 10.3171/2015.1.JNS141301. Epub 2015 Aug 28. PMID 26315004
- [Background] Miskin N, Patel H, Franceschi AM, Ades-Aron B, Le A, Damadian BE, Stanton C, Serulle Y, Golomb J, Gonen O, Rusinek H, George AE; Alzheimer's Disease Neuroimaging Initiative. Diagnosis of Normal-Pressure Hydrocephalus: Use of Traditional Measures in the Era of Volumetric MR Imaging. Radiology. 2017 Oct;285(1):197-205. doi: 10.1148/radiol.2017161216. Epub 2017 May 10. PMID 28498794
- [Background] Neikter J, Agerskov S, Hellstrom P, Tullberg M, Starck G, Ziegelitz D, Farahmand D. Ventricular Volume Is More Strongly Associated with Clinical Improvement Than the Evans Index after Shunting in Idiopathic Normal Pressure Hydrocephalus. AJNR Am J Neuroradiol. 2020 Jul;41(7):1187-1192. doi: 10.3174/ajnr.A6620. Epub 2020 Jun 11. PMID 32527841
- [Background] Hakim S, Adams RD. The special clinical problem of symptomatic hydrocephalus with normal cerebrospinal fluid pressure. Observations on cerebrospinal fluid hydrodynamics. J Neurol Sci. 1965 Jul-Aug;2(4):307-27. doi: 10.1016/0022-510x(65)90016-x. No abstract available. PMID 5889177